CLINICAL TRIAL: NCT06463067
Title: Evaluation Of The Effects Of Reading Educational Books, Showing Videos, And Playing Mobile Games On Dental Anxiety In Children
Brief Title: Books, Videos And Mobile Games İn Pediatric Dentistry
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Melek Belevcikli, Assistant professor, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bülent Ecevit Üniversitesi
Record Dates: First submitted 2024-05-17; First posted 2024-06-17 (Actual); Last update posted 2024-06-17 (Actual); Status verified 2024-06

CONDITIONS: Dental Anxiety; Child, Only
Keywords: book; Dental anxiety; Behavior management; video; mobil game

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Play group (Other): Before the examination process, the child was asked to select one of the five faces on the Facial Image Scale. The dentist evaluated and scored the patient's behaviors based on the categories in the Frankl Behavior Scale. Parents were asked to answer the questions in the Corah Dental Anxiety Scale on behalf of their children to assess their dental anxiety, and results were scored. Subsequently, the children's heart rate was measured and recorded with a pulse oximeter attached to the index finger of the left hand. Prior to the examination procedure, The patients in Play Group played a mobile game called 'Dentist' before the examination. After that patients were examined, and their anxiety levels were assessed using the same methods following the examination procedure
  Interventions: Behavioral: playing mobile game
- Book group (Other): Before the examination, the child was asked to choose one of five faces from the Facial Image Scale. The dentist assessed and scored the patient's behaviour using the Frankl Behaviour Scale. Parents were asked to complete the Corah Dental Anxiety Scale on behalf of their children to assess their dental anxiety and the results were scored. The children's heart rate was then measured and recorded using a pulse oximeter attached to the index finger of the left hand. The researcher then read the storybook "Elif Goes to the Dentist" and showed the children pictures of dental instruments as described in the book. Behavioural techniques were used to examine the patients, and their anxiety levels were assessed after the examination using the same methods.
  Interventions: Behavioral: reading book
- Video group (Other): Before the examination, the child was asked to choose one of the five faces on the Facial Image Scale. The dentist assessed the patient's behaviour using the Frankl Behaviour Scale. Parents were asked to answer the questions on the Corah Dental Anxiety Scale on behalf of their children to assess their dental anxiety, and the results were scored. The children's heart rate was then measured and recorded using a pulse oximeter attached to the index finger of the left hand. Patients in the video group then watched an animated video entitled 'First meeting with the dentist' before the examination, and dental instruments were introduced using the terminology mentioned in the video. Using behavioural techniques, the patients were examined and their anxiety levels were assessed using the same methods after the examination.
  Interventions: Behavioral: watching video
- Tell-show-do group (Other): Before the examination, the child was asked to choose one of five faces on the Facial Image Scale (FIS). The dentist assessed and scored the patient's behaviour using the Frankl Behaviour Scale. Parents were asked to complete the Corah Dental Anxiety Scale on behalf of their children to assess their dental anxiety, and the results were scored. The children's heart rate was then measured and recorded using a pulse oximeter attached to the index finger of the left hand. Following the application of the behavioural techniques, the patients were examined and their anxiety levels were assessed using the same methods after the examination procedure.
  Interventions: Behavioral: tell-show-do group

INTERVENTIONS:
Behavioral: playing mobile game — Changes in anxiety levels were measured by playing a mobile game to children before dental examination.
  Arms: Play group
Behavioral: reading book — Changes in anxiety levels were measured by reading books to children before dental examination.
  Arms: Book group
Behavioral: watching video — Changes in anxiety levels were measured by showing a video to children before dental examination.
  Arms: Video group
Behavioral: tell-show-do group — Before the dental examination, the tell-show-do technique was applied to the children and the changes in their anxiety levels were measured.
  Arms: Tell-show-do group

SUMMARY:
The objective of this study was to examine the impact of educational video viewing, reading educational books, and playing educational mobile games on children's dental anxiety prior to dental examinations. The main questions it aims to answer are:

1. Does reading educational books before dental examinations reduce dental anxiety in children?
2. Does watching educational videos before dental examinations reduce children's dental anxiety?
3. Does playing educational mobile games before dental check-ups reduce dental anxiety in children?

DETAILED DESCRIPTION:
ackground: Behaviour management techniques have an important place in paediatric dentistry. However, alternative methods may be needed if they are found to be ineffective in reducing children's dental anxiety.Aim: This study aimed to evaluate the impact of reading educational books, watching videos and playing mobile games from the child's, dentist's and parent's perspective on children's dental anxiety before treatment.

Methods: A total of 160 patients were randomly assigned to four groups. Anxiety levels of patients in each group were assessed using the Facial Image Scale, the Frankl Behaviour Scale and pulse oximetry. The Corah Dental Anxiety Scale was administered to parents to assess their child's anxiety level. The first group was exposed to the tell-show-do technique, the second group read a book, the third group watched a video and the fourth group played a mobile phone game. The children in each group were then assessed. Anxiety levels were then reassessed using the same scales.

ELIGIBILITY:
Inclusion Criteria:

1. The child must be between 3-6 years old
2. No previous dentist experience
3. No systemic disease or syndrome

Exclusion Criteria:

1. The child is under 3 years old and over 6 years old
2. Having been to the dentist before for an examination or dental treatment.
3. Having any systemic disease or syndrome

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
anxiety level according to the child | after dental examination to 10 minute
  We evaluated the effects of reading informative books, playing mobile games and watching videos after the dental examination on dental anxiety by measuring the Facial Image Scale (In the facial image scale consisting of 5 different faces, the happiest face is given a value of 1 while the unhappiest face is given a value of 5 and scoring is done according to the face chosen by the children.)

SECONDARY OUTCOMES:
child's anxiety level according to the researcher | after dental examination to 30 minute
  We evaluated the effects of reading informative books, playing mobile games and watching videos after the dental examination on dental anxiety by measuring the Frankl Behaviour Scale, (Frankl Behavior Scale: is based on the observation, evaluation and scoring of the child's behavior by the dentist. In this scale, which is filled in by the dentist, the child's behavior in different situations is classified as strongly negative (1), negative (2), positive (3), strongly positive (4). )

OTHER OUTCOMES:
child's level of dental anxiety from the parents' perspective | after dental examination to 24 hour
  We evaluated the effects of reading informative books, playing mobile games and watching videos after the dental examination on dental anxiety by measuring the Corah Dental Anxiety Scale (Corah Dental Anxiety Scale: It consists of four short questions designed to measure dental anxiety levels related to dental treatments. Each question has 5 answers and the answers are scored from 1 to 5 by the physician. A score of less than 13 indicates a low level of anxiety, 13-14 indicates a moderate level of anxiety, and 15 and above indicates a high level of anxiety. If the child is too young to understand the questions, the questions can be answered by the parent or caregiver.)
children's anxiety levels according to heart rate | after dental examination to 2 minute
  We evaluated the effects of reading informative books, playing mobile games and watching videos after the dental examination on dental anxiety by measuring the heart rate (It has been reported that pulse rate measurement is a reliable method for determining anxiety level. Increased anxiety level leads to increased heart rate.It has been reported that pulse rate measurement is a reliable method for determining the level of anxiety. Increased anxiety level leads to increased heart rate. Pulse rates of 80-120 between 2-4 years of age and 75-115 between 4-6 years of age are considered normal in children.)

CONTACTS AND LOCATIONS:
Overall Officials: gamze kılıç, 1, Principal Investigator — Bulent Ecevit University
Locations (1):
- Bülent Ecevit Univercity, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No